CLINICAL TRIAL: NCT05914675
Title: Efficacy and Safety of Letermovir for Primary Prophylaxis of Cytomegalovirus Infection After HLA-haploidentical Hematopoietic Stem Cell Transplantation
Brief Title: Letermovir for Primary Prophylaxis of Cytomegalovirus Infection After R+HID-HSCT
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT-CMV-PP-01
Record Dates: First submitted 2023-06-13; First posted 2023-06-22 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-05

CONDITIONS: The Incidence of Peripheral Blood CMV Activation and Confirmed Clinically Significant CMV Infection Within 24 Weeks After Transplantation
Keywords: CMV reactivation; CMV infection; HSCT
MeSH Terms: conditions — Cytomegalovirus Infections | interventions — letermovir

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- treatment arm (Experimental)
  Interventions: Drug: Letermovir

INTERVENTIONS:
Drug: Letermovir — For enrolled patients, Letermovir would be administered at a dose of 480 mg per day (or 240 mg per day in patients taking cyclosporine). The regimen would start between +7~+14d after transplantation. The total duration of dosing was approximately 100 days or 14 weeks.

SUMMARY:
To evaluate the efficacy and safety of primary prophylaxis of CMV reactivation, clinically significant CMV infection with oral letermovir in Chinese R+ haplo-HSCT patients, as well as treatment-related mortality and all-cause mortality within 24 weeks after transplantation. For enrolled patients, Letermovir would be administered at a dose of 480 mg per day (or 240 mg per day in patients taking cyclosporine). The regimen would start between +7~+14d after transplantation. The total duration of dosing was approximately 100 days or 14 weeks.

ELIGIBILITY:
Inclusion Criteria:

* (1) Underwent HLA-haploidentical donor HSCT and could receive investigational drug within 28 days of transplantation. (2) have documented seropositivity for CMV (recipient CMV IgG seropositivity [R+]) within 1 year before HSCT., plasma CMV-DNA copy number less than the lower limit of detection within 5 days before enrollment (threshold of 1000 copies/ml in our hospital); (3) Age elder than or equal to 18 years; (4) Informed consent may be signed by themselves. (5) HIV negative, HBV, HCV negative; (6) Informed consent must be signed before the start of the study procedures, and informed consent must be signed by the patient himself or his immediate family. Considering the patient 's condition, if the patient' s signature is unfavorable for disease treatment, the informed consent form should be signed by the legal guardian or the patient 's immediate family member.

Exclusion Criteria:

* Subjects who met any of the following criteria were not enrolled in this study: (1) received a previous allogeneic HSCT; (2) has a history of CMV end-organ disease within 6 months prior to enrollment, or has evidence of CMV viremia from a central or local laboratory at any time prior to enrollment; (3) received within 7 days prior to screening or plans to receive during the study any of the following: ganciclovir, valganciclovir, foscarnet sodium, acyclovir (daily oral dose > 3200 mg, or daily intravenous dose > 25 mg/kg), valacyclovir (daily oral dose > 3000 mg), famciclovir (daily oral dose > 1500 mg); (4) received within 30 days prior to screening or plans to receive during the study any of the following: cidofovir, CMV high-titer gamma globulin, any investigational anti-CMV therapy or biological agent; (5) has severe hepatic insufficiency (defined as Child-Pugh Class C; (6) has serum aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 5 xthe upper limit of normal (ULN) or serum total bilirubin > 2.5 x ULN.(7) has end-stage renal impairment with a creatinine clearance less than 10 mL/min. (8) has both moderate hepatic insufficiency AND moderate renal insufficiency; (9) Uncontrolled infection at enrollment; (10) requires mechanical ventilation or is hemodynamically unstable at the time of enrollment; (11) has documented positive results for human immunodeficiency virus antibody (HIVAb), hepatitis C virus antibody (HCV-Ab) with detectable HCV RNA, or hepatitis B surface antigen (HBsAg) within 90 days prior to randomization (12) has active solid tumor malignancies with the exception of localized basal cell or squamous cell skin cancer or the condition under treatment (e.g., lymphomas). (13) Suffering from mental disorders or other conditions and unable to cooperate with the requirements of study treatment and monitoring; 14) unable or unwilling to sign the consent form; 15) pregnant or lactating women; 16) patients with other special conditions assessed as unqualified by the investigator.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
CMV reactivation or clinically significant CMV infection incidence | 24 weeks after HSCT
  The incidence of peripheral blood cytomegalovirus activation and confirmed clinically significant CMV infection

IPD SHARING:
Plan to Share IPD: No